CLINICAL TRIAL: NCT04108468
Title: An Investigator-initiated Double-blind, Parallel-group Randomised Controlled Trial of GOLimumab and Methotrexate Versus Methotrexate in Very Early PsA Using Clinical and Whole Body MRI Outcomes: the GOLMePsA Study.
Brief Title: GOLimumab and Methotrexate Versus Methotrexate in Very Early PsA
Acronym: GOLMePsA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: The Leeds Teaching Hospitals NHS Trust (Other)
Collaborators: Janssen Pharmaceutica N.V., Belgium (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RR13/10782; 14/EM/0124 (Other: Research Ethics Committee)
Record Dates: First submitted 2019-09-26; First posted 2019-09-30 (Actual); Results first posted 2025-12-02 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Psoriatic Arthritis
MeSH Terms: conditions — Arthritis, Psoriatic | interventions — Methotrexate; golimumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Methotrexate (Active Comparator)
  Interventions: Drug: Methotrexate
- Golimumab & Methotrexate (Experimental)
  Interventions: Drug: Methotrexate; Drug: Golimumab

INTERVENTIONS:
Drug: Methotrexate — Methotrexate
Drug: Golimumab — Simponi
  Arms: Golimumab & Methotrexate

SUMMARY:
An investigator-initiated double-blind, parallel-group randomised controlled trial of Methotrexate versus GOLimumab and Methotrexate in very early PsA using clinical and whole body MRI outcomes.

DETAILED DESCRIPTION:
Phase IIIb. Early Psoriatic Arthritis. Investigator initiated, double-blind, randomized, placebo-controlled, two-armed, parallel-group, single centre trial.

The Primary Objective is to assess whether the combination of golimumab with methotrexate and steroids is superior to standard care (MTX monotherapy plus steroids) in reducing clinical disease activity in patients with early, treatment naïve PsA.

ELIGIBILITY:
Inclusion Criteria:

Male and female patients aged ≥18 years at the time of signing the Informed Consent Form.

Subjects with a diagnosis of psoriatic arthritis as per the Classification for Psoriatic Arthritis (CASPAR) criteria (Appendix 4) confirmed less than 24 months prior to screening.

Subjects with active PsA defined as the presence of at least 3/68 tender and at least 3/66 swollen joints or 2 swollen and 2 tender joints plus one affected entheseal site (Achilles tendon and/or plantar fascia) at baseline.

Are treatment naïve to DMARDs. Are capable of understanding and signing an informed consent form. Women of childbearing potential or men capable of fathering children must be using adequate birth control measures (eg, abstinence, oral contraceptives, intrauterine device, barrier method with spermicide, surgical sterilization) during the study and for 6 months after receiving the last administration of study agent. Female subjects of childbearing potential must test negative for pregnancy. Female subjects must agree to not donate eggs (ova, oocytes) during the study and for 6 months after last dose of study agent. Male subjects must agree to not donate sperm while in the study and for 6 months after last dose of study agent.

Patients fulfilling the following TB criteria:

7.1. Have no history of latent or active TB prior to screening. An exception is made for subjects with a history of latent TB and documentation of having completed appropriate treatment for latent TB 3 years prior to the first administration of study agent. It is the responsibility of the investigator to verify the adequacy of previous antituberculous treatment and provide appropriate documentation.

7.2. Have no signs or symptoms suggestive of active TB upon medical history and/or physical examination.

7.3. Have had no close contact with a person with active TB or, if there has been such a contact, will be referred to a physician specializing in TB to undergo additional evaluation, and if warranted, receive appropriate treatment as if having latent TB prior to or simultaneously with the first administration of study agent.

7.4. Within 6 weeks prior to the administration of study agent, either have a negative QuantiFERON-TB Gold test result or have a newly identified positive QuantiFERON-TB Gold test result in which active TB has been ruled out and for which appropriate treatment for latent TB has been initiated either prior to or simultaneously with the first administration of study agent.

7.5. In the event of 2 indeterminate QuantiFERON-TB Gold in-tube tests results, the subjects will be treated as if having latent TB prior or simultaneously with the first administration of study agent.

7.6. Have a chest radiograph (posterior-anterior view), read by a qualified radiologist, whose diagnostic assessment is consistent with no evidence of current active TB or old inactive TB, and taken within 12 months of the study.

7.7. Have a screening laboratory test result as follows: 7.7.1. Hb≥8.5 g/dL or ≥5.3 mmol/L 7.7.2. White blood cell (WBC) count ≥3.5x103 cells/uL 7.7.3. Neutrophils ≥1.5 x103 cells/uL 7.7.4. Platelets ≥100x103 cells/uL 7.7.5. Serum alanine aminotransferase (ALT) and aspartate aminotransferase (AST) levels not exceeding 1.5 times the upper limit of normal (UKN) for the central laboratory conducting the test.

7.7.6. Serum creatinine not exceeding 1.5 mg/dL

Exclusion Criteria:

1. Received previous treatment with any DMARDs.
2. Received previous treatment with golimumab or other tumour necrosis factor inhibitor (TNFi) or other biologic drugs.
3. Any chronic inflammatory arthritis diagnosed before 16 years old. Exclusions for general safety

Patients with significant concurrent medical diseases including uncompensated congestive heart failure, myocardial infarction within 52 weeks from screening, unstable angina pectoris, uncontrolled hypertension (BP>160/95), severe pulmonary disease, or history of human immunodeficiency virus (HIV) infection, immunodeficiency syndromes, central nervous system (CNS) demyelinating events suggestive of multiple sclerosis, renal or gastrointestinal conditions, which in the opinion of the investigator places the patient at an unacceptable risk for participation in the study or would make implementation of the protocol difficult.

Patients with cancer or a history of cancer (other than resected cutaneous basal cell carcinoma, and in situ cervical cancer) within 5 years of screening.

Patients with current crystal or infective arthritis. Patients with chronic infection of the upper respiratory tract (eg. Sinusitis), chest (eg. Bronchiectatic lung disease), urinary tract or skin (eg. Paronychia, chronic ulcers, open wounds) within 4 weeks of screening.

Patients who have a chest radiograph within 3 months prior to the first administration of study agent that shows an abnormality suggestive of a malignancy or current active infection, including TB, histoplasmosis or coccidioidomycosis.

Patients with any ongoing or active infection or any major episode of infection requiring hospitalization or treatment with IV antibiotics within the preceding 30 days of screening and/or orally administered antibiotics in the preceding 15 days of screening.

Patients with abnormal liver function including known liver cirrhosis, fibrosis, or known alcoholic steatohepatitis (NASH) at the time of screening or abnormal blood tests as shown by:

Aminotransferase (AST) / alanine aminotransferase (ALT) > 3x ULN, OR Bilirubin >51umol/L

Patients with known severe hypoproteinaemia at the time of screening, e.g. in nephrotic syndrome or impaired renal function, as shown by:

• Serum Creatinine > 133 mol/L

Patients with known significantly impaired bone marrow function as for example significant anaemia, leukopaenia, neutropaenia or thrombocytopaenia as shown by the following laboratory values at the time of screening:

White blood cells < 3000 x 106/L Platelets < 125 x 109/L Haemoglobin < 9.0 g/dL for males and < 8.5 g/dL for females Patients with a history of latent or active TB prior to screening will not be eligible. For exceptions refer to inclusion criteria.

Subjects must undergo screening for hepatitis B virus (HBV). At a minimum, this includes testing for HBsAg (surface antigen), anti-HBs (surface antibody), and anti-HBc total (core antibody total).

11.1. Subjects who test positive for surface antigen (HBsAg+) are not eligible for this study, regardless of the results of other hepatitis B tests.

11.2. Subjects who test negative for surface antibody (HBsAg-) and test positive for core antibody (anti-HBc+) and surface antibody (anti-HBs+) are eligible for this study.

11.3. Subjects who test positive only for surface antibody (anti-HBs+) are eligible for this study.

11.4. Subjects who test positive only for core antibody (anti-HBc+) must undergo further testing for hepatitis B deoxyribonucleic acid (HBV DNA test). If the HBV DNA test is positive, the subject is not eligible for this study. If the HBV DNA test is negative, the subject is eligible for this study. In the event the DNA test cannot be performed, the subject is not eligible for the study.

Primary or secondary immunodeficiency (history of or currently active) unless related to primary disease under investigation.

Pregnancy, lactation (nursing) or women of child-bearing potential (WCBP) unwilling to use an effective birth control measure (Appendix 1) whilst receiving treatment and after the last dose of protocol treatment as indicated in the relevant SmPC/IB.

Men whose partners are of child-bearing potential but who are unwilling to use an effective birth control measure whilst receiving treatment and after the last dose of protocol treatment as indicated in the relevant SmPC/IB.

Patients who have received any corticosteroids within 4 weeks prior to screening.

Patients with a history of confirmed blood dyscrasia. Patients with a history of mental illness that would interfere with their ability to comply with the study protocol.

Patients with a history of drug and/or alcohol abuse that would interfere with their ability to comply with the study protocol.

Patients with a history of any viral hepatitis within 1 year of screening Patients who have received or are expected to receive any live virus or bacterial vaccinations or treatments that include live organisms (eg. a therapeutic infectious agent such as BCG that is instilled into the bladder for the treatment of cancer) within 3 months prior to the first administration of study agent, during the trial, or within 6 months after the last administration of the study agent.

Patients who demonstrate Hypersensitivity to the active substance, or any of the excipients detailed in the SmPC.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2015-10-27 (Actual); Primary Completion 2023-07 (Actual); Study Completion 2023-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- The Leeds Teaching Hospitals NHS Trust, Leeds, West Yorkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Methotrexate | Golimumab & Methotrexate
Started | 41 | 43
Completed | 38 | 39
Not Completed | 3 | 4
Not completed — Physician Decision | 0 | 1
Not completed — Lost to Follow-up | 0 | 1
Not completed — Non-compliance | 1 | 1
Not completed — Unable to attend final visit | 2 | 0
Not completed — Missed study medication | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Methotrexate | Golimumab & Methotrexate | Total
Number analyzed (Participants) | 41 | 43 | 84
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 39 | 40 | 79
  >=65 years | 2 | 3 | 5
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.9 (12.5) | 42.1 (12.5) | 42.5 (12.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 19 | 38
  Male | 22 | 24 | 46
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 32 | 29 | 61
  Asian | 2 | 3 | 5
  Other | 1 | 1 | 2
  Not stated | 6 | 10 | 16
Region of Enrollment [Number; unit: participants]
  United Kingdom | 41 | 43 | 84
PASDAS [Mean (Standard Deviation); unit: units on a scale] — The Psoriatic Arthritis Disease Activity Score (PASDAS) is a composite outcome based on the physician global VAS, participant global VAS, SF-36 physical component score, 66 swollen joint count, 68 tender joint count, Leeds enthesitis index, tender dactylitis count and C-reactive protein. The PASDAS ranges from 0-10, with higher values indicating higher disease activity.
  units on a scale | 5.6 (1.1) | 5.9 (1.3) | 5.7 (1.2)
Leeds Enthesitis Index [Mean (Standard Deviation); unit: score on a scale] — The Leeds Enthesitis Index is a count of the number of tender entheses out of a possible 6 (lateral epicondyle, left and right, medial femoral condyle, left and right, Achilles tendon insertion, left and right). A higher score indicates a wider extent of enthesitis.
  score on a scale | 1.51 (1.76) | 1.37 (1.47) | 1.44 (1.62)
Leeds Dactylitis Index [Mean (Standard Deviation); unit: units on a scale] — The Leeds Dactylitis Index measures dactylitis severity. The ratio of the circumference of the affected digit to the circumference of the digit on the opposite side is measured. Each dactylitic digit is defined by a minimum increase of 10% in circumference over the contra-lateral digit. The calculated ratio is then multiplied by a tenderness score of 0 (non-tender), 1 (tender), 2 (tender and wince) or 3 (tender and withdraw). Tenderness is assessed in the area between the joints. The results of each digit are then added to produce a total score. Range 0-~40, higher score means worse dactylitis
  units on a scale | 26.60 (30.56) | 38.04 (50.85) | 32.45 (42.32)
Psoriatic Arthritis Skin Index Score [Median (Inter-Quartile Range); unit: units on a scale] — The PASI combines assessments of the extent of body-surface involvement in 4 anatomical regions (head, trunk, arms, and legs) and the severity of desquamation, erythema, and plaque induration/infiltration (thickness) in each region, yielding an overall score of 0 for no Pso to 72 for the most severe disease.
  units on a scale | 2.6 [0.9 to 5.1] | 3.4 [0.5 to 6.9] | 2.7 [0.6 to 6.0]
Modified Nail Psoriasis Severity Index (mNAPSI) [Mean (Standard Deviation); unit: units on a scale] — Each fingernail is scored for the presence and the severity of pitting, onycholysis, oil-drop dyschromia and nail plate crumbling (score 0-3) and the presence or absence of splinter haemorrhages, leuconychia, red spots in the lunula and nail bed hyperkeratosis (score 1 for each if present). The scale ranges from 0 to 140, higher scores indicate worse nail psoriasis.
  units on a scale | 7.25 (11.26) | 11.36 (18.15) | 9.35 (15.23)
Composite Psoriatic Disease Activity Index (CPDAI) [Mean (Standard Deviation); unit: units on a scale] — Domains include peripheral arthritis (assessed by 68 tender joints count, 66 swollen joints count, and the Health Assessment Questionnaire), skin as assessed by the PASI and the DLQI, enthesitis as assessed by the number of sites with enthesitis and the HAQ, dactylitis as assessed by the number of digits affected, and spinal disease as assessed by the BASDAI and ASQoL. Scores range from 0 to 15. Higher scores indicate higher disease activity.
  units on a scale | 6.4 (2.7) | 7.0 (2.6) | 6.7 (2.6)
Ultrasound Global OMERACT-EULAR System Score (GLOESS) [Mean (Standard Deviation); unit: units on a scale] — Joints are scored 0-3 for grey scale and power Doppler; a combined score takes a value of 0 if grey scale=0, if grey scale is >0 then the combined score is the maximum of the grey scale and power Doppler scores. Scores for individual joints are then summated to give a total global score. For the set of joints scanned in all participants, this ranges from 0-72; for the subset in whom a wider set of joints were scanned, this ranges from 0 to 144. Higher scores indicate worse synovial hypertrophy and vascularisation.
  units on a scale | 21.6 (11.2) | 24.8 (13.0) | 23.2 (12.2)
Ultrasound Entheseal Inflammatory Score [Mean (Standard Deviation); unit: units on a scale] — Grey scale changes in the entheses related to inflammation (entheseal hypoechogenicity and thickening) are added to power Doppler scores. The score ranges from 0-70, higher scores indicate worse entheseal inflammation.
  units on a scale | 4.2 (3.7) | 5.4 (3.9) | 4.8 (3.8)
Ultrasound Entheseal Chronicity Score [Mean (Standard Deviation); unit: units on a scale] — Grey scale changes related to chronic findings (calcifications, erosion and enthesophytes) are summated. The score ranges from 0-50; higher scores indicate a greater extent of chronic entheseal pathology.
  units on a scale | 3.0 (3.1) | 3.5 (3.0) | 3.2 (3.0)
Participant Disease Activity Visual Analogue Scale [Mean (Standard Deviation); unit: units on a scale] — Participants are asked to assess their current level of joint pain by marking a vertical line on a 100 mm horizontal VAS where 0 represents no joint pain ("excellent") and 100 represents worst imaginable joint pain ("poor").
  units on a scale | 52.1 (25.2) | 59.1 (21.4) | 55.7 (23.5)
Dermatology Life Quality Index (DLQI) [Median (Inter-Quartile Range); unit: units on a scale] — The DLQI is a simple, patient administered, 10 question, validated, quality of life questionnaire that covers 6 domains including symptoms and feelings, daily activities, leisure, work and school, personal relationships and treatment. Response categories include "not at all", "a lot" and "very much" with corresponding scores of 1, 2 and 3 respectively and unanswered ("not relevant") responses scored as "0". Totals range from 0 to 30 (less to more impairment) and a 5-point change from baseline is considered clinically relevant.
  units on a scale | 3.0 [1.0 to 7.0] | 5.0 [1.0 to 9.0] | 3.5 [1.0 to 8.5]
36-Item Short Form Health Survey (SF-36) Physical Component Summary [Mean (Standard Deviation); unit: units on a scale] — The SF-36 physical component summary scale ranges from 0-100, with scores above 50 indicating better than average physical health.
  units on a scale | 37.5 (9.9) | 32.5 (10.0) | 34.9 (10.2)
36-Item Short Form Health Survey (SF-36) Mental Component Summary [Mean (Standard Deviation); unit: units on a scale] — The SF-36 mental component summary scale ranges from 0-100, with scores above 50 indicating better than average mental health.
  units on a scale | 46.6 (12.5) | 46.7 (10.7) | 46.7 (11.5)

OUTCOME MEASURES:

1. Primary Outcome: Psoriatic Arthritis Disease Activity Score (PASDAS) at 24 Weeks
Description: The Psoriatic Arthritis Disease Activity Score ranges from 0-10; higher scores represent a worse outcome.
Time Frame: 24 weeks
Population: Full analysis set
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Methotrexate | Golimumab & Methotrexate
Number analyzed (Participants) | 41 | 43
score on a scale | 3.09 (1.32) | 2.70 (1.38)
Statistical Analysis 1: Comparison: Methotrexate vs Golimumab & Methotrexate; Test type: Superiority; p = 0.064, Regression, Linear; Adjusted for baseline PASDAS and poly/oligoarthritis status (the stratification variable). Multiple imputation addressed missing data; Mean Difference (Final Values) = -0.55, 95% CI 2-sided [-1.12 to 0.03] — The mean difference was adjusted pre-specified covariates, and calculated following multiple imputation. The individual group means reported were unadjusted, available case estimates. The placebo/methotrexate arm was the reference category

2. Secondary Outcome: Psoriatic Arthritis Disease Activity Score (PASDAS) at 12 Weeks.
Description: The Psoriatic Arthritis Disease Activity Score ranges from 0-10; higher scores represent a worse outcome.
Time Frame: 12 weeks
Population: Full analysis set
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Methotrexate | Golimumab & Methotrexate
Number analyzed (Participants) | 41 | 43
score on a scale | 3.70 (1.62) | 3.01 (1.31)
Statistical Analysis 1: Comparison: Methotrexate vs Golimumab & Methotrexate; Test type: Superiority; p = 0.007, Regression, Linear; Adjusted for baseline BASDAS and poly/oligoarthritis status (the stratification variable). Multiple imputation addressed missing data; Mean Difference (Final Values) = -0.86, 95% CI 2-sided [-1.48 to -0.24] — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: Psoriatic Arthritis Disease Activity Score (PASDAS) at 36 Weeks.
Description: The Psoriatic Arthritis Disease Activity Score ranges from 0-10; higher scores represent a worse outcome.
Time Frame: 36 weeks
Population: Full analysis set
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Methotrexate | Golimumab & Methotrexate
Number analyzed (Participants) | 41 | 43
score on a scale | 3.30 (1.70) | 2.93 (3.42)
Statistical Analysis 1: Comparison: Methotrexate vs Golimumab & Methotrexate; Test type: Superiority; p = 0.096, Regression, Linear; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.58, 95% CI 2-sided [-1.26 to 0.11] — [estimate comment as in outcome 1, analysis 1]

4. Secondary Outcome: Psoriatic Arthritis Disease Activity Score (PASDAS) at 52 Weeks.
Description: The Psoriatic Arthritis Disease Activity Score ranges from 0-10; higher scores represent a worse outcome.
Time Frame: 52 weeks
Population: Full analysis set
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Methotrexate | Golimumab & Methotrexate
Number analyzed (Participants) | 41 | 43
score on a scale | 3.36 (1.39) | 3.42 (1.55)
Statistical Analysis 1: Comparison: Methotrexate vs Golimumab & Methotrexate; Test type: Superiority; p = 0.844, Regression, Linear; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.07, 95% CI 2-sided [-0.72 to 0.59] — [estimate comment as in outcome 1, analysis 1]

5. Secondary Outcome: Composite Psoriatic Disease Activity Index (CPDAI) at 12 Weeks.
Description: The Composite Psoriatic Disease Activity Index ranges from 0-15; higher scores represent a worse outcome.
Time Frame: 12 weeks
Population: Full analysis set
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Methotrexate | Golimumab & Methotrexate
Number analyzed (Participants) | 41 | 43
score on a scale | 4.10 (2.76) | 3.49 (2.41)
Statistical Analysis 1: Comparison: Methotrexate vs Golimumab & Methotrexate; Test type: Superiority; p = 0.041, Regression, Linear; Adjusted for baseline CPDAI and poly/oligoarthritis status (the stratification variable). Multiple imputation addressed missing data; Mean Difference (Final Values) = -0.96, 95% CI 2-sided [-1.88 to -0.04] — [estimate comment as in outcome 1, analysis 1]

6. Secondary Outcome: Composite Psoriatic Disease Activity Index (CPDAI) at 24 Weeks.
Description: The Composite Psoriatic Disease Activity Index ranges from 0-15; higher scores represent a worse outcome.
Time Frame: 24 weeks
Population: Full analysis set
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Methotrexate | Golimumab & Methotrexate
Number analyzed (Participants) | 41 | 43
score on a scale | 3.24 (2.58) | 3.12 (2.45)
Statistical Analysis 1: Comparison: Methotrexate vs Golimumab & Methotrexate; Test type: Superiority; p = 0.375, Regression, Linear; [statistical method as in outcome 5, analysis 1]; Mean Difference (Final Values) = -0.44, 95% CI 2-sided [-1.41 to 0.54] — [estimate comment as in outcome 1, analysis 1]

7. Secondary Outcome: Composite Psoriatic Disease Activity Index (CPDAI) at 36 Weeks.
Description: The Composite Psoriatic Disease Activity Index ranges from 0-15; higher scores represent a worse outcome.
Time Frame: 36 weeks
Population: Full analysis set
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Methotrexate | Golimumab & Methotrexate
Number analyzed (Participants) | 41 | 43
score on a scale | 2.97 (2.69) | 3.17 (2.80)
Statistical Analysis 1: Comparison: Methotrexate vs Golimumab & Methotrexate; Test type: Superiority; p = 0.392, Regression, Linear; [statistical method as in outcome 5, analysis 1]; Mean Difference (Final Values) = -0.44, 95% CI 2-sided [-1.46 to 0.58] — [estimate comment as in outcome 1, analysis 1]

8. Secondary Outcome: Composite Psoriatic Disease Activity Index (CPDAI) at 52 Weeks.
Description: The Composite Psoriatic Disease Activity Index ranges from 0-15; higher scores represent a worse outcome.
Time Frame: 52 weeks
Population: Full analysis set
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Methotrexate | Golimumab & Methotrexate
Number analyzed (Participants) | 41 | 43
score on a scale | 3.03 (2.71) | 3.49 (2.75)
Statistical Analysis 1: Comparison: Methotrexate vs Golimumab & Methotrexate; Test type: Superiority; p = 0.541, Regression, Linear; [statistical method as in outcome 5, analysis 1]; Mean Difference (Final Values) = -0.32, 95% CI 2-sided [-1.34 to 0.71] — [estimate comment as in outcome 1, analysis 1]

9. Secondary Outcome: Participant Disease Activity Visual Analogue Score at 24 Weeks.
Description: The Participant Disease Activity Visual Analogue Score ranges from 0-100; higher scores represent a worse outcome.
Time Frame: 24 weeks
Population: Full analysis set
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Methotrexate | Golimumab & Methotrexate
Number analyzed (Participants) | 41 | 43
score on a scale | 27.56 (23.54) | 27.72 (23.42)
Statistical Analysis 1: Comparison: Methotrexate vs Golimumab & Methotrexate; Test type: Superiority; p = 0.633, Regression, Linear; Adjusted for baseline score and poly/oligoarthritis status (the stratification variable). Multiple imputation addressed missing data; Mean Difference (Final Values) = -2.35, 95% CI 2-sided [-12.14 to 7.43] — [estimate comment as in outcome 1, analysis 1]

10. Secondary Outcome: Participant Disease Activity Visual Analogue Score at 52 Weeks.
Description: The Participant Disease Activity Visual Analogue Score ranges from 0-100; higher scores represent a worse outcome.
Time Frame: 52 weeks
Population: Full analysis set
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Methotrexate | Golimumab & Methotrexate
Number analyzed (Participants) | 41 | 43
score on a scale | 32.73 (25.62) | 36.57 (26.06)
Statistical Analysis 1: Comparison: Methotrexate vs Golimumab & Methotrexate; Test type: Superiority; p = 0.826, Regression, Linear; [statistical method as in outcome 9, analysis 1]; Mean Difference (Final Values) = 1.24, 95% CI 2-sided [-9.95 to 12.43] — [estimate comment as in outcome 1, analysis 1]

11. Secondary Outcome: 36-item Short Form Health Survey (SF-36) Physical Component Score at 24 Weeks.
Description: The 36-item Short Form Health Survey (SF-36) Physical Component Score ranges from 0-100; higher scores represent a better outcome.
Time Frame: 24 weeks
Population: Full analysis set
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Methotrexate | Golimumab & Methotrexate
Number analyzed (Participants) | 41 | 43
score on a scale | 45.62 (9.45) | 46.10 (9.32)
Statistical Analysis 1: Comparison: Methotrexate vs Golimumab & Methotrexate; Test type: Superiority; p = 0.268, Regression, Linear; [statistical method as in outcome 9, analysis 1]; Mean Difference (Final Values) = 2.24, 95% CI 2-sided [-1.76 to 6.25] — [estimate comment as in outcome 1, analysis 1]

12. Secondary Outcome: 36-item Short Form Health Survey (SF-36) Physical Component Score at 52 Weeks.
Description: as for outcome 11
Time Frame: 52 weeks
Population: Full analysis set
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Methotrexate | Golimumab & Methotrexate
Number analyzed (Participants) | 41 | 43
score on a scale | 44.44 (10.25) | 42.80 (10.38)
Statistical Analysis 1: Comparison: Methotrexate vs Golimumab & Methotrexate; Test type: Superiority; p = 0.605, Regression, Linear; [statistical method as in outcome 9, analysis 1]; Mean Difference (Final Values) = 1.21, 95% CI 2-sided [-3.42 to 5.83] — [estimate comment as in outcome 1, analysis 1]

13. Secondary Outcome: 36-item Short Form Health Survey (SF-36) Mental Component Score at 24 Weeks.
Description: The 36-item Short Form Health Survey (SF-36) Mental Component Score ranges from 0-100; higher scores represent a better outcome.
Time Frame: 24 weeks
Population: Full analysis set
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Methotrexate | Golimumab & Methotrexate
Number analyzed (Participants) | 41 | 43
score on a scale | 52.11 (9.34) | 51.27 (8.84)
Statistical Analysis 1: Comparison: Methotrexate vs Golimumab & Methotrexate; Test type: Superiority; p = 0.620, Regression, Linear; [statistical method as in outcome 9, analysis 1]; Mean Difference (Final Values) = -0.85, 95% CI 2-sided [-4.23 to 2.54] — [estimate comment as in outcome 1, analysis 1]

14. Secondary Outcome: 36-item Short Form Health Survey (SF-36) Mental Component Score at 52 Weeks.
Description: as for outcome 13
Time Frame: 52 weeks
Population: Full analysis set
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Methotrexate | Golimumab & Methotrexate
Number analyzed (Participants) | 41 | 43
score on a scale | 52.44 (10.03) | 51.65 (9.75)
Statistical Analysis 1: Comparison: Methotrexate vs Golimumab & Methotrexate; Test type: Superiority; p = 0.449, Regression, Linear; [statistical method as in outcome 9, analysis 1]; Mean Difference (Final Values) = -1.39, 95% CI 2-sided [-5.02 to 2.24] — [estimate comment as in outcome 1, analysis 1]

15. Secondary Outcome: Ultrasound Global OMERACT-EULAR System Score (GLOESS) at 12 Weeks.
Description: In the joint set scanned in the Full Analysis Set, the Ultrasound Global OMERACT-EULAR System Score ranged from 0-72; higher scores represent a worse outcome.
Time Frame: 12 weeks
Population: Full analysis set
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Methotrexate | Golimumab & Methotrexate
Number analyzed (Participants) | 41 | 43
score on a scale | 18.74 (10.12) | 23.07 (11.74)
Statistical Analysis 1: Comparison: Methotrexate; Test type: Superiority; p = 0.364, Regression, Linear; [statistical method as in outcome 9, analysis 1]; Mean Difference (Final Values) = 1.72, 95% CI 2-sided [-2.04 to 5.48] — [estimate comment as in outcome 1, analysis 1]

16. Secondary Outcome: Ultrasound Global OMERACT-EULAR System Score (GLOESS) at 24 Weeks.
Description: as for outcome 15
Time Frame: 24 weeks
Population: Full analysis set
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Methotrexate | Golimumab & Methotrexate
Number analyzed (Participants) | 41 | 43
score on a scale | 20.63 (10.06) | 22.44 (10.26)
Statistical Analysis 1: Comparison: Methotrexate vs Golimumab & Methotrexate; Test type: Superiority; p = 0.806, Regression, Linear; [statistical method as in outcome 9, analysis 1]; Mean Difference (Final Values) = 0.51, 95% CI 2-sided [-3.60 to 4.61] — [estimate comment as in outcome 1, analysis 1]

17. Secondary Outcome: Ultrasound Global OMERACT-EULAR System Score (GLOESS) at 36 Weeks.
Description: as for outcome 15
Time Frame: 36 weeks
Population: Full analysis set
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Methotrexate | Golimumab & Methotrexate
Number analyzed (Participants) | 41 | 43
score on a scale | 22.46 (9.83) | 24.20 (7.96)
Statistical Analysis 1: Comparison: Methotrexate vs Golimumab & Methotrexate; Test type: Superiority; p = 0.588, Regression, Linear; [statistical method as in outcome 9, analysis 1]; Mean Difference (Final Values) = 1.05, 95% CI 2-sided [-2.79 to 4.89] — [estimate comment as in outcome 1, analysis 1]

18. Secondary Outcome: Ultrasound Entheseal Inflammatory Score at 12 Weeks.
Description: The Ultrasound Entheseal Inflammatory Score ranged from 0-70; a higher score represents a worse outcome.
Time Frame: 12 weeks
Population: Full analysis set
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Methotrexate | Golimumab & Methotrexate
Number analyzed (Participants) | 41 | 43
score on a scale | 4.86 (4.80) | 4.68 (4.28)
Statistical Analysis 1: Comparison: Methotrexate vs Golimumab & Methotrexate; Test type: Superiority; p = 0.372, Regression, Linear; [statistical method as in outcome 9, analysis 1]; Mean Difference (Final Values) = -0.76, 95% CI 2-sided [-2.45 to 0.93] — [estimate comment as in outcome 1, analysis 1]

19. Secondary Outcome: Ultrasound Entheseal Inflammatory Score at 24 Weeks.
Description: The Ultrasound Entheseal Inflammatory Score ranged from 0-70; a higher score represents a worse outcome.
Time Frame: 24 weeks
Population: Full analysis set
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Methotrexate | Golimumab & Methotrexate
Number analyzed (Participants) | 41 | 43
score on a scale | 4.89 (4.49) | 4.90 (3.92)
Statistical Analysis 1: Comparison: Methotrexate vs Golimumab & Methotrexate; Test type: Superiority; p = 0.781, Regression, Linear; [statistical method as in outcome 9, analysis 1]; Mean Difference (Final Values) = -0.25, 95% CI 2-sided [-2.05 to 1.55] — [estimate comment as in outcome 1, analysis 1]

20. Secondary Outcome: Ultrasound Entheseal Inflammatory Score at 36 Weeks.
Description: The Ultrasound Entheseal Inflammatory Score ranged from 0-70; a higher score represents a worse outcome.
Time Frame: 36 weeks
Population: Full analysis set
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Methotrexate | Golimumab & Methotrexate
Number analyzed (Participants) | 41 | 43
score on a scale | 6.17 (6.49) | 4.14 (3.45)
Statistical Analysis 1: Comparison: Methotrexate vs Golimumab & Methotrexate; Test type: Superiority; p = 0.037, Regression, Linear; [statistical method as in outcome 9, analysis 1]; Mean Difference (Final Values) = -2.26, 95% CI 2-sided [-4.39 to -0.14] — [estimate comment as in outcome 1, analysis 1]

21. Secondary Outcome: Ultrasound Entheseal Chronicity Score at 12 Weeks.
Description: The Ultrasound Entheseal Chronicity Score ranged from 0-50; a higher score represents a worse outcome.
Time Frame: 12 weeks
Population: Full analysis set
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Methotrexate | Golimumab & Methotrexate
Number analyzed (Participants) | 41 | 43
score on a scale | 3.17 (2.38) | 2.50 (2.79)
Statistical Analysis 1: Comparison: Methotrexate vs Golimumab & Methotrexate; Test type: Superiority; p = 0.058, Regression, Linear; [statistical method as in outcome 9, analysis 1]; Mean Difference (Final Values) = -0.95, 95% CI 2-sided [-1.93 to 0.03] — [estimate comment as in outcome 1, analysis 1]

22. Secondary Outcome: Ultrasound Entheseal Chronicity Score at 24 Weeks.
Description: The Ultrasound Entheseal Chronicity Score ranged from 0-50; a higher score represents a worse outcome.
Time Frame: 24 weeks
Population: Full analysis set
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Methotrexate | Golimumab & Methotrexate
Number analyzed (Participants) | 41 | 43
score on a scale | 2.85 (2.31) | 2.63 (2.21)
Statistical Analysis 1: Comparison: Methotrexate vs Golimumab & Methotrexate; Test type: Superiority; p = 0.213, Regression, Linear; [statistical method as in outcome 9, analysis 1]; Mean Difference (Final Values) = -0.60, 95% CI 2-sided [-1.54 to 0.35] — [estimate comment as in outcome 1, analysis 1]

23. Secondary Outcome: Ultrasound Entheseal Chronicity Score at 36 Weeks.
Description: The Ultrasound Entheseal Chronicity Score ranged from 0-50; a higher score represents a worse outcome.
Time Frame: 36 weeks
Population: Full analysis set
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Methotrexate | Golimumab & Methotrexate
Number analyzed (Participants) | 41 | 43
score on a scale | 2.79 (2.64) | 2.97 (2.66)
Statistical Analysis 1: Comparison: Methotrexate vs Golimumab & Methotrexate; Test type: Superiority; p = 0.606, Regression, Linear; [statistical method as in outcome 9, analysis 1]; Mean Difference (Final Values) = 0.31, 95% CI 2-sided [-0.88 to 1.50] — [estimate comment as in outcome 1, analysis 1]

24. Secondary Outcome: Leeds Enthesitis Index at 12 Weeks
Description: The Leeds Enthesitis Index ranges from 0-6; a higher score represents a worse outcome.
Time Frame: 12 Weeks
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Methotrexate | Golimumab & Methotrexate
Number analyzed (Participants) | 41 | 43
score on a scale | 0.95 (1.76) | 0.74 (1.35)
Statistical Analysis 1: Comparison: Methotrexate vs Golimumab & Methotrexate; Test type: Superiority; p = 0.971, Negative binomial regression; [statistical method as in outcome 9, analysis 1]; Incidence-rate ratio = 1.01, 95% CI 2-sided [0.48 to 2.14] — The placebo/methotrexate arm was the reference category

25. Secondary Outcome: Leeds Enthesitis Index at 24 Weeks
Description: The Leeds Enthesitis Index ranges from 0-6; a higher score represents a worse outcome.
Time Frame: 24 Weeks
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Methotrexate | Golimumab & Methotrexate
Number analyzed (Participants) | 41 | 43
score on a scale | 0.61 (1.34) | 0.53 (0.98)
Statistical Analysis 1: Comparison: Methotrexate vs Golimumab & Methotrexate; Test type: Superiority; p = 0.817, Negative binomial regression; [statistical method as in outcome 9, analysis 1]; Incidence-rate ratio = 1.10, 95% CI 2-sided [0.49 to 2.46] — The placebo/methotrexate group was the reference category

26. Secondary Outcome: Leeds Enthesitis Index at 36 Weeks
Description: The Leeds Enthesitis Index ranges from 0-6; a higher score represents a worse outcome.
Time Frame: 36 Weeks
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Methotrexate | Golimumab & Methotrexate
Number analyzed (Participants) | 41 | 43
score on a scale | 0.65 (1.37) | 0.74 (1.43)
Statistical Analysis 1: Comparison: Methotrexate vs Golimumab & Methotrexate; Test type: Superiority; p = 0.441, Negative binomial regression; [statistical method as in outcome 9, analysis 1]; Incidence-rate ratio = 1.35, 95% CI 2-sided [0.63 to 2.93] — The placebo/methotrexate group was the reference category

27. Secondary Outcome: Leeds Enthesitis Index at 52 Weeks
Description: The Leeds Enthesitis Index ranges from 0-6; a higher score represents a worse outcome.
Time Frame: 52 Weeks
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Methotrexate | Golimumab & Methotrexate
Number analyzed (Participants) | 41 | 43
score on a scale | 0.43 (1.09) | 0.50 (0.97)
Statistical Analysis 1: Comparison: Methotrexate vs Golimumab & Methotrexate; Test type: Superiority; p = 0.563, Negative binomial regression; [statistical method as in outcome 9, analysis 1]; Incidence-rate ratio = 1.29, 95% CI 2-sided [0.55 to 3.03] — The placebo/methotrexate group was the reference category

28. Secondary Outcome: Leeds Dactylitis Index at 12 Weeks
Description: The Leeds Dactylitis Index ranges from 0-~40; a higher score represents a worse outcome.
Time Frame: 12 Weeks
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Methotrexate | Golimumab & Methotrexate
Number analyzed (Participants) | 41 | 43
units on a scale | 11.46 (19.88) | 2.22 (7.92)
Statistical Analysis 1: Comparison: Methotrexate vs Golimumab & Methotrexate; Test type: Superiority; p = 0.083, Negative binomial regression; [statistical method as in outcome 9, analysis 1]; Incidence-rate ratio = 0.17, 95% CI 2-sided [0.02 to 1.26] — The placebo/methotrexate group was the reference category

29. Secondary Outcome: Leeds Dactylitis Index at 24 Weeks
Description: The Leeds Dactylitis Index ranges from 0-~40; a higher score represents a worse outcome.
Time Frame: 24 Weeks
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Methotrexate | Golimumab & Methotrexate
Number analyzed (Participants) | 41 | 43
units on a scale | 5.04 (17.10) | 0.48 (2.52)
Statistical Analysis 1: Comparison: Methotrexate vs Golimumab & Methotrexate; Test type: Superiority; p = 0.432, Negative binomial regression; [statistical method as in outcome 9, analysis 1]; Incidence-rate ratio = 0.26, 95% CI 2-sided [0.01 to 7.64] — The placebo/methotrexate group was the reference category

30. Secondary Outcome: Leeds Dactylitis Index at 36 Weeks
Description: The Leeds Dactylitis Index ranges from 0-~40; a higher score represents a worse outcome.
Time Frame: 36 Weeks
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Methotrexate | Golimumab & Methotrexate
Number analyzed (Participants) | 41 | 43
units on a scale | 4.38 (11.31) | 3.36 (15.15)
Statistical Analysis 1: Comparison: Methotrexate vs Golimumab & Methotrexate; Test type: Superiority; p = 0.071, Negative binomial regression; [statistical method as in outcome 9, analysis 1]; Incidence-rate ratio = 0.11, 95% CI 2-sided [0.01 to 1.21] — The placebo/methotrexate group was the reference category

31. Secondary Outcome: Leeds Dactylitis Index at 52 Weeks
Description: The Leeds Dactylitis Index ranges from 0-~40; a higher score represents a worse outcome.
Time Frame: 52 Weeks
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Methotrexate | Golimumab & Methotrexate
Number analyzed (Participants) | 41 | 43
units on a scale | 6.58 (14.89) | 3.45 (14.76)
Statistical Analysis 1: Comparison: Methotrexate vs Golimumab & Methotrexate; Test type: Superiority; p = 0.037, Negative binomial regression; [statistical method as in outcome 9, analysis 1]; Incidence-rate ratio = 0.06, 95% CI 2-sided [0.00 to 0.84] — The placebo/methotrexate group was the reference category

32. Secondary Outcome: The Modified Nail Psoriasis Severity Index (mNAPSI) at 12 Weeks
Description: The Modified Nail Psoriasis Severity Index ranges from 0-140; a higher score represents a worse outcome.
Time Frame: 12 Weeks
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Methotrexate | Golimumab & Methotrexate
Number analyzed (Participants) | 41 | 43
units on a scale | 4.78 (8.73) | 6.37 (10.66)
Statistical Analysis 1: Comparison: Methotrexate vs Golimumab & Methotrexate; Test type: Superiority; p = 0.296, Negative binomial regression; [statistical method as in outcome 9, analysis 1]; Incidence-rate ratio = 0.68, 95% CI 2-sided [0.32 to 1.41] — The placebo/methotrexate group was the reference category

33. Secondary Outcome: The Modified Nail Psoriasis Severity Index (mNAPSI) at 24 Weeks
Description: The Modified Nail Psoriasis Severity Index ranges from 0-140; a higher score represents a worse outcome.
Time Frame: 24 Weeks
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Methotrexate | Golimumab & Methotrexate
Number analyzed (Participants) | 41 | 43
units on a scale | 4.02 (6.41) | 3.12 (6.88)
Statistical Analysis 1: Comparison: Methotrexate vs Golimumab & Methotrexate; Test type: Superiority; p = 0.081, Negative binomial regression; [statistical method as in outcome 9, analysis 1]; Incidence-rate ratio = 0.51, 95% CI 2-sided [0.23 to 1.09] — The placebo/methotrexate group was the reference category

34. Secondary Outcome: The Modified Nail Psoriasis Severity Index (mNAPSI) at 36 Weeks
Description: The Modified Nail Psoriasis Severity Index ranges from 0-140; a higher score represents a worse outcome.
Time Frame: 36 Weeks
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Methotrexate | Golimumab & Methotrexate
Number analyzed (Participants) | 41 | 43
units on a scale | 4.47 (7.73) | 5.50 (11.16)
Statistical Analysis 1: Comparison: Methotrexate vs Golimumab & Methotrexate; Test type: Superiority; p = 0.458, Negative binomial regression; [statistical method as in outcome 9, analysis 1]; Incidence-rate ratio = 0.75, 95% CI 2-sided [0.36 to 1.59] — The placebo/methotrexate group was the reference category

35. Secondary Outcome: The Modified Nail Psoriasis Severity Index (mNAPSI) at 52 Weeks
Description: The Modified Nail Psoriasis Severity Index ranges from 0-140; a higher score represents a worse outcome.
Time Frame: 52 Weeks
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Methotrexate | Golimumab & Methotrexate
Number analyzed (Participants) | 41 | 43
units on a scale | 3.91 (7.32) | 7.72 (12.27)
Statistical Analysis 1: Comparison: Methotrexate vs Golimumab & Methotrexate; Test type: Superiority; p = 0.798, Negative binomial regression; [statistical method as in outcome 9, analysis 1]; Incidence-rate ratio = 1.12, 95% CI 2-sided [0.46 to 2.72] — The placebo/methotrexate group was the reference category

36. Secondary Outcome: Psoriasis Area and Severity Index (PASI) Score at 12 Weeks
Description: The Psoriasis Area and Severity Index ranges from 0-72; a higher score represents a worse outcome.
Time Frame: 12 Weeks
Population: Full Analysis Set
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Methotrexate | Golimumab & Methotrexate
Number analyzed (Participants) | 41 | 43
score on a scale | 1.00 [0.00 to 2.10] | 0.20 [0.00 to 1.20]
Statistical Analysis 1: Comparison: Methotrexate vs Golimumab & Methotrexate; Test type: Superiority; p = 0.512, Quantile (median) regression; [statistical method as in outcome 9, analysis 1]; Median Difference (Final Values) = -0.38, 95% CI 2-sided [-1.53 to 0.77] — The placebo/methotrexate group was the reference category

37. Secondary Outcome: Psoriasis Area and Severity Index (PASI) Score at 24 Weeks
Description: The Psoriasis Area and Severity Index ranges from 0-72; a higher score represents a worse outcome.
Time Frame: 24 Weeks
Population: Full Analysis Set
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Methotrexate | Golimumab & Methotrexate
Number analyzed (Participants) | 41 | 43
score on a scale | 0.60 [0.00 to 1.60] | 0.00 [0.00 to 0.70]
Statistical Analysis 1: Comparison: Methotrexate vs Golimumab & Methotrexate; Test type: Superiority; p = 0.320, Quantile (median) regression; [statistical method as in outcome 9, analysis 1]; Median Difference (Final Values) = -0.44, 95% CI 2-sided [-1.33 to 0.44] — The placebo/methotrexate group was the reference category

38. Secondary Outcome: Psoriasis Area and Severity Index (PASI) Score at 36 Weeks
Description: The Psoriasis Area and Severity Index ranges from 0-72; a higher score represents a worse outcome.
Time Frame: 36 Weeks
Population: Full Analysis Set
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Methotrexate | Golimumab & Methotrexate
Number analyzed (Participants) | 41 | 43
score on a scale | 0.70 [0.00 to 1.75] | 0.00 [0.00 to 0.60]
Statistical Analysis 1: Comparison: Methotrexate vs Golimumab & Methotrexate; Test type: Superiority; p = 0.220, Quantile (median) regression; [statistical method as in outcome 9, analysis 1]; Median Difference (Final Values) = -0.47, 95% CI 2-sided [-1.22 to 0.28] — The placebo/methotrexate group was the reference category

39. Secondary Outcome: Psoriasis Area and Severity Index (PASI) Score at 52 Weeks
Description: The Psoriasis Area and Severity Index ranges from 0-72; a higher score represents a worse outcome.
Time Frame: 52 Weeks
Population: Full Analysis Set
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Methotrexate | Golimumab & Methotrexate
Number analyzed (Participants) | 41 | 43
score on a scale | 0.40 [0.00 to 1.60] | 0.55 [0.00 to 1.80]
Statistical Analysis 1: Comparison: Methotrexate vs Golimumab & Methotrexate; Test type: Superiority; p = 0.912, Quantile (median) regression; [statistical method as in outcome 9, analysis 1]; Median Difference (Final Values) = 0.05, 95% CI 2-sided [-0.85 to 0.95] — The placebo/methotrexate group was the reference category

40. Secondary Outcome: Dermatology Life Quality Index (DLQI) Score at 24 Weeks
Description: The Dermatology Life Quality Index ranges from 0-30; a higher score represents a worse outcome.
Time Frame: 24 Weeks
Population: Full Analysis Set
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Methotrexate | Golimumab & Methotrexate
Number analyzed (Participants) | 41 | 43
score on a scale | 1.00 [0.00 to 2.00] | 1.00 [0.00 to 1.00]
Statistical Analysis 1: Comparison: Methotrexate vs Golimumab & Methotrexate; Test type: Superiority; p = 0.281, Quantile (median) regression; [statistical method as in outcome 9, analysis 1]; Median Difference (Final Values) = -0.50, 95% CI 2-sided [-1.42 to 0.42] — The placebo/methotrexate group was the reference category

41. Secondary Outcome: Dermatology Life Quality Index (DLQI) Score at 52 Weeks
Description: The Dermatology Life Quality Index ranges from 0-30; a higher score represents a worse outcome.
Time Frame: 52 Weeks
Population: Full Analysis Set
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Methotrexate | Golimumab & Methotrexate
Number analyzed (Participants) | 41 | 43
score on a scale | 1.00 [0.00 to 2.00] | 1.00 [0.00 to 4.00]
Statistical Analysis 1: Comparison: Methotrexate vs Golimumab & Methotrexate; Test type: Superiority; p = 0.985, Quantile (median) regression; [statistical method as in outcome 9, analysis 1]; Median Difference (Final Values) = 0.01, 95% CI 2-sided [-1.44 to 1.47] — The placebo/methotrexate group was the reference category

42. Secondary Outcome: Minimal Disease Activity (MDA) at 12 Weeks
Description: Minimal Disease Activity (coded 0=No, 1=Yes) is achieved when at least 5 of the 7 following criteria are met: Tender joint count (/68) ≤1 Swollen joint count (/66) ≤1 PASI ≤1 or BSA≤3 Patient pain VAS ≤15 Patient global disease activity VAS ≤20 HAQ ≤0.5 Enthesitis count ≤1.
Time Frame: 12 Weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Methotrexate | Golimumab & Methotrexate
Number analyzed (Participants) | 41 | 43
Participants | 18 | 20
Statistical Analysis 1: Comparison: Methotrexate vs Golimumab & Methotrexate; Test type: Superiority; p = 0.869, Regression, Logistic; Adjusted for poly/oligoarthritis status (the stratification variable). Multiple imputation addressed missing data; Odds Ratio (OR) = 1.08, 95% CI 2-sided [0.45 to 2.60] — The placebo/methotrexate group was the reference category

43. Secondary Outcome: Minimal Disease Activity (MDA) at 24 Weeks
Description: as for outcome 42
Time Frame: 24 Weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Methotrexate | Golimumab & Methotrexate
Number analyzed (Participants) | 41 | 43
Participants | 24 | 24
Statistical Analysis 1: Comparison: Methotrexate vs Golimumab & Methotrexate; Test type: Superiority; p = 0.802, Regression, Logistic; Adjusted for poly/oligoarthritis status (the stratification variable). Multiple imputation addressed missing data; Odds Ratio (OR) = 0.90, 95% CI 2-sided [0.38 to 2.13] — The placebo/methotrexate group was the reference category

44. Secondary Outcome: Minimal Disease Activity (MDA) at 36 Weeks
Description: as for outcome 42
Time Frame: 36 Weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Methotrexate | Golimumab & Methotrexate
Number analyzed (Participants) | 41 | 43
Participants | 22 | 25
Statistical Analysis 1: Comparison: Methotrexate vs Golimumab & Methotrexate; Test type: Superiority; p = 0.767, Regression, Logistic; Adjusted for poly/oligoarthritis status (the stratification variable). Multiple imputation addressed missing data; Odds Ratio (OR) = 1.14, 95% CI 2-sided [0.48 to 2.72] — The placebo/methotrexate group was the reference category

45. Secondary Outcome: Minimal Disease Activity (MDA) at 52 Weeks
Description: as for outcome 42
Time Frame: 52 Weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Methotrexate | Golimumab & Methotrexate
Number analyzed (Participants) | 41 | 43
Participants | 20 | 17
Statistical Analysis 1: Comparison: Methotrexate vs Golimumab & Methotrexate; Test type: Superiority; p = 0.315, Regression, Logistic; Adjusted for poly/oligoarthritis status (the stratification variable). Multiple imputation addressed missing data; Odds Ratio (OR) = 0.63, 95% CI 2-sided [0.26 to 1.55] — The placebo/methotrexate group was the reference category

46. Secondary Outcome: American College of Rheumatology 20 (ACR20) Response at 12 Weeks
Description: American College of Rheumatology 20 Response (coded 0=No, 1=Yes) is achieved when there is:
  * 20% improvement in both TJC (68 joints count) and SJC (66 joints count) and
  * 20% improvement in at least 3 of the following 5 ACR Core set criteria:
    1. Patient's Assessment of Pain Visual Analogue Scale (VAS)
    2. Patient's Global Assessment of Disease Activity VAS
    3. Physician's Global Assessment of Disease Activity VAS
    4. Patient's Assessment of Physical Function as measured by the HAQ-DI
    5. Acute phase reactant as measured by CRP
Time Frame: 12 Weeks
Population: Full Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Methotrexate | Golimumab & Methotrexate
Number analyzed (Participants) | 41 | 43
Participants | 23 | 28
Statistical Analysis 1: Comparison: Methotrexate vs Golimumab & Methotrexate; Test type: Superiority; p = 0.516, Regression, Logistic; Adjusted for poly/oligoarthritis status (the stratification variable). Multiple imputation addressed missing data; Odds Ratio (OR) = 1.34, 95% CI 2-sided [0.55 to 3.27] — The placebo/methotrexate group was the reference category

47. Secondary Outcome: American College of Rheumatology 20 (ACR20) Response at 24 Weeks
Description: as for outcome 46
Time Frame: 24 Weeks
Population: Full Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Methotrexate | Golimumab & Methotrexate
Number analyzed (Participants) | 41 | 43
Participants | 27 | 28
Statistical Analysis 1: Comparison: Methotrexate vs Golimumab & Methotrexate; Test type: Superiority; p = 0.939, Regression, Logistic; Adjusted for poly/oligoarthritis status (the stratification variable). Multiple imputation addressed missing data; Odds Ratio (OR) = 0.97, 95% CI 2-sided [0.39 to 2.38] — The placebo/methotrexate group was the reference category

48. Secondary Outcome: American College of Rheumatology 20 (ACR20) Response at 36 Weeks
Description: as for outcome 46
Time Frame: 36 Weeks
Population: Full Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Methotrexate | Golimumab & Methotrexate
Number analyzed (Participants) | 41 | 43
Participants | 24 | 27
Statistical Analysis 1: Comparison: Methotrexate vs Golimumab & Methotrexate; Test type: Superiority; p = 0.701, Regression, Logistic; Adjusted for poly/oligoarthritis status (the stratification variable). Multiple imputation addressed missing data; Odds Ratio (OR) = 1.19, 95% CI 2-sided [0.48 to 2.94] — The placebo/methotrexate group was the reference category

49. Secondary Outcome: American College of Rheumatology 20 (ACR20) Response at 52 Weeks
Description: as for outcome 46
Time Frame: 52 Weeks
Population: Full Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Methotrexate | Golimumab & Methotrexate
Number analyzed (Participants) | 41 | 43
Participants | 28 | 23
Statistical Analysis 1: Comparison: Methotrexate vs Golimumab & Methotrexate; Test type: Superiority; p = 0.124, Regression, Logistic; Adjusted for poly/oligoarthritis status (the stratification variable). Multiple imputation addressed missing data; Odds Ratio (OR) = 0.48, 95% CI 2-sided [0.19 to 1.22] — The placebo/methotrexate group was the reference category

50. Secondary Outcome: American College of Rheumatology 50 (ACR50) Response at 12 Weeks
Description: American College of Rheumatology 50 Response (coded 0=No, 1=Yes) is achieved when there is:
  * 50% improvement in both TJC (68 joints count) and SJC (66 joints count) and
  * 50% improvement in at least 3 of the following 5 ACR Core set criteria:
    1. Patient's Assessment of Pain Visual Analogue Scale (VAS)
    2. Patient's Global Assessment of Disease Activity VAS
    3. Physician's Global Assessment of Disease Activity VAS
    4. Patient's Assessment of Physical Function as measured by the HAQ-DI
    5. Acute phase reactant as measured by CRP
Time Frame: 12 Weeks
Population: Full Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Methotrexate | Golimumab & Methotrexate
Number analyzed (Participants) | 41 | 43
Participants | 12 | 20
Statistical Analysis 1: Comparison: Methotrexate vs Golimumab & Methotrexate; Test type: Superiority; p = 0.161, Regression, Logistic; Adjusted for poly/oligoarthritis status (the stratification variable). Multiple imputation addressed missing data; Odds Ratio (OR) = 1.89, 95% CI 2-sided [0.78 to 4.63] — The placebo/methotrexate group was the reference category

51. Secondary Outcome: American College of Rheumatology 50 (ACR50) Response at 24 Weeks
Description: as for outcome 50
Time Frame: 24 Weeks
Population: Full Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Methotrexate | Golimumab & Methotrexate
Number analyzed (Participants) | 41 | 43
Participants | 15 | 21
Statistical Analysis 1: Comparison: Methotrexate vs Golimumab & Methotrexate; Test type: Superiority; p = 0.251, Regression, Logistic; Adjusted for poly/oligoarthritis status (the stratification variable). Multiple imputation addressed missing data; Odds Ratio (OR) = 1.67, 95% CI 2-sided [0.70 to 4.02] — The placebo/methotrexate group was the reference category

52. Secondary Outcome: American College of Rheumatology 50 (ACR50) Response at 36 Weeks
Description: as for outcome 50
Time Frame: 36 Weeks
Population: Full Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Methotrexate | Golimumab & Methotrexate
Number analyzed (Participants) | 41 | 43
Participants | 16 | 21
Statistical Analysis 1: Comparison: Methotrexate vs Golimumab & Methotrexate; Test type: Superiority; p = 0.363, Regression, Logistic; Adjusted for poly/oligoarthritis status (the stratification variable). Multiple imputation addressed missing data; Odds Ratio (OR) = 1.50, 95% CI 2-sided [0.63 to 3.60] — The placebo/methotrexate group was the reference category

53. Secondary Outcome: American College of Rheumatology 50 (ACR50) Response at 52 Weeks
Description: as for outcome 50
Time Frame: 52 Weeks
Population: Full Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Methotrexate | Golimumab & Methotrexate
Number analyzed (Participants) | 41 | 43
Participants | 15 | 16
Statistical Analysis 1: Comparison: Methotrexate vs Golimumab & Methotrexate; Test type: Superiority; p = 0.991, Regression, Logistic; Adjusted for poly/oligoarthritis status (the stratification variable). Multiple imputation addressed missing data; Odds Ratio (OR) = 0.99, 95% CI 2-sided [0.40 to 2.46] — The placebo/methotrexate group was the reference category

54. Secondary Outcome: American College of Rheumatology 70 (ACR70) Response at 12 Weeks
Description: American College of Rheumatology 70 Response (coded 0=No, 1=Yes) is achieved when there is:
  * 70% improvement in both TJC (68 joints count) and SJC (66 joints count) and
  * 70% improvement in at least 3 of the following 5 ACR Core set criteria:
    1. Patient's Assessment of Pain Visual Analogue Scale (VAS)
    2. Patient's Global Assessment of Disease Activity VAS
    3. Physician's Global Assessment of Disease Activity VAS
    4. Patient's Assessment of Physical Function as measured by the HAQ-DI
    5. Acute phase reactant as measured by CRP
Time Frame: 12 Weeks
Population: Full Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Methotrexate | Golimumab & Methotrexate
Number analyzed (Participants) | 41 | 43
Participants | 6 | 15
Statistical Analysis 1: Comparison: Methotrexate vs Golimumab & Methotrexate; Test type: Superiority; p = 0.037, Regression, Logistic; Adjusted for poly/oligoarthritis status (the stratification variable). Multiple imputation addressed missing data; Odds Ratio (OR) = 3.12, 95% CI 2-sided [1.07 to 9.10] — The placebo/methotrexate group was the reference category

55. Secondary Outcome: American College of Rheumatology 70 (ACR70) Response at 24 Weeks
Description: as for outcome 54
Time Frame: 24 Weeks
Population: Full Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Methotrexate | Golimumab & Methotrexate
Number analyzed (Participants) | 41 | 43
Participants | 10 | 19
Statistical Analysis 1: Comparison: Methotrexate vs Golimumab & Methotrexate; Test type: Superiority; p = 0.056, Regression, Logistic; Odds Ratio (OR) = 2.50, 95% CI 2-sided [0.98 to 6.40] — The placebo/methotrexate group was the reference category

56. Secondary Outcome: American College of Rheumatology 70 (ACR70) Response at 36 Weeks
Description: as for outcome 54
Time Frame: 36 Weeks
Population: Full Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Methotrexate | Golimumab & Methotrexate
Number analyzed (Participants) | 41 | 43
Participants | 9 | 14
Statistical Analysis 1: Comparison: Methotrexate vs Golimumab & Methotrexate; Test type: Superiority; p = 0.277, Regression, Logistic; Adjusted for poly/oligoarthritis status (the stratification variable). Multiple imputation addressed missing data; Odds Ratio (OR) = 1.72, 95% CI 2-sided [0.65 to 4.57] — The placebo/methotrexate group was the reference category

57. Secondary Outcome: American College of Rheumatology 70 (ACR70) Response at 52 Weeks
Description: as for outcome 54
Time Frame: 52 Weeks
Population: Full Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Methotrexate | Golimumab & Methotrexate
Number analyzed (Participants) | 41 | 43
Participants | 8 | 11
Statistical Analysis 1: Comparison: Methotrexate vs Golimumab & Methotrexate; Test type: Superiority; p = 0.548, Regression, Logistic; Adjusted for poly/oligoarthritis status (the stratification variable). Multiple imputation addressed missing data; Odds Ratio (OR) = 1.38, 95% CI 2-sided [0.48 to 3.92] — The placebo/methotrexate group was the reference category

58. Secondary Outcome: Psoriatic Arthritis Response Criteria (PsARC) Response at 12 Weeks
Description: Psoriatic Arthritis Response Criteria Response (coded 0=No, 1=Yes) is defined by improvement from baseline assessment in 2 of 4 criteria, 1 of which must be a joint count; there must not be worsening in any of the 4 criteria:
  1. At least 30% reduction in tender joint grade (total of 68 joints graded 0-3)
  2. At least 30% reduction in swollen joint grade (total of 66 joints graded 0-3)
  3. At least a 1 point reduction in physician's assessment of articular disease (1-5 Likert scale)
  4. At least a 1 point reduction in patient's assessment of articular disease (1-5 Likert scale)
Time Frame: 12 Weeks
Population: Full Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Methotrexate | Golimumab & Methotrexate
Number analyzed (Participants) | 41 | 43
Participants | 26 | 37
Statistical Analysis 1: Comparison: Methotrexate vs Golimumab & Methotrexate; Test type: Superiority; p = 0.018, Regression, Logistic; Adjusted for poly/oligoarthritis status (the stratification variable). Multiple imputation addressed missing data; Odds Ratio (OR) = 3.70, 95% CI 2-sided [1.25 to 10.97] — The placebo/methotrexate group was the reference category

59. Secondary Outcome: Psoriatic Arthritis Response Criteria (PsARC) Response at 24 Weeks
Description: as for outcome 58
Time Frame: 24 Weeks
Population: Full Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Methotrexate | Golimumab & Methotrexate
Number analyzed (Participants) | 41 | 43
Participants | 36 | 38
Statistical Analysis 1: Comparison: Methotrexate vs Golimumab & Methotrexate; Test type: Superiority; p = 0.926, Regression, Logistic; Adjusted for poly/oligoarthritis status (the stratification variable). Multiple imputation addressed missing data; Odds Ratio (OR) = 1.06, 95% CI 2-sided [0.28 to 4.02] — The placebo/methotrexate group was the reference category

60. Secondary Outcome: Psoriatic Arthritis Response Criteria (PsARC) Response at 36 Weeks
Description: as for outcome 58
Time Frame: 36 Weeks
Population: Full Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Methotrexate | Golimumab & Methotrexate
Number analyzed (Participants) | 41 | 43
Participants | 33 | 38
Statistical Analysis 1: Comparison: Methotrexate vs Golimumab & Methotrexate; Test type: Superiority; p = 0.385, Regression, Logistic; Adjusted for poly/oligoarthritis status (the stratification variable). Multiple imputation addressed missing data; Odds Ratio (OR) = 1.73, 95% CI 2-sided [0.50 to 5.94] — The placebo/methotrexate group was the reference category

61. Secondary Outcome: Psoriatic Arthritis Response Criteria (PsARC) Response at 52 Weeks
Description: as for outcome 58
Time Frame: 52 Weeks
Population: Full Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Methotrexate | Golimumab & Methotrexate
Number analyzed (Participants) | 41 | 43
Participants | 27 | 28
Statistical Analysis 1: Comparison: Methotrexate vs Golimumab & Methotrexate; Test type: Superiority; p = 0.684, Regression, Logistic; Adjusted for poly/oligoarthritis status (the stratification variable). Multiple imputation addressed missing data; Odds Ratio (OR) = 0.82, 95% CI 2-sided [0.32 to 2.12] — The placebo/methotrexate group was the reference category

62. Secondary Outcome: Psoriatic Arthritis Skin Index (PASI) Response at 12 Weeks
Description: Psoriatic Arthritis Skin Index (PASI) Response (coded 0=No, 1=Yes) is defined as an improvement of at least 75% in the PASI compared to baseline.
Time Frame: 12 Weeks
Population: Full Analysis Set (restricted to those with >=3% body surface area affected by psoriasis at baseline)
Measure: Count of Participants; unit: Participants
Arm/Group | Methotrexate | Golimumab & Methotrexate
Number analyzed (Participants) | 8 | 13
Participants | 0 | 7
Statistical Analysis 1: Comparison: Methotrexate vs Golimumab & Methotrexate; Test type: Superiority; p = 0.063, Regression, Logistic; Adjusted for poly/oligoarthritis status (the stratification variable). Multiple imputation addressed missing data; Odds Ratio (OR) = 16.72, 95% CI 2-sided [0.86 to 326.19] — The placebo/methotrexate group was the reference category

63. Secondary Outcome: Psoriatic Arthritis Skin Index (PASI) Response at 24 Weeks
Description: as for outcome 62
Time Frame: 24 Weeks
Population: Full Analysis Set (restricted to those with >=3% body surface area affected by psoriasis at baseline)
Measure: Count of Participants; unit: Participants
Arm/Group | Methotrexate | Golimumab & Methotrexate
Number analyzed (Participants) | 8 | 13
Participants | 3 | 11
Statistical Analysis 1: Comparison: Methotrexate vs Golimumab & Methotrexate; Test type: Superiority; p = 0.041, Regression, Logistic; Adjusted for poly/oligoarthritis status (the stratification variable). Multiple imputation addressed missing data; Odds Ratio (OR) = 8.90, 95% CI 2-sided [1.09 to 72.42] — The placebo/methotrexate group was the reference category

64. Secondary Outcome: Psoriatic Arthritis Skin Index (PASI) Response at 36 Weeks
Description: as for outcome 62
Time Frame: 36 Weeks
Population: Full Analysis Set (restricted to those with >=3% body surface area affected by psoriasis at baseline)
Measure: Count of Participants; unit: Participants
Arm/Group | Methotrexate | Golimumab & Methotrexate
Number analyzed (Participants) | 8 | 13
Participants | 2 | 9
Statistical Analysis 1: Comparison: Methotrexate vs Golimumab & Methotrexate; Test type: Superiority; p = 0.069, Regression, Logistic; Adjusted for poly/oligoarthritis status (the stratification variable). Multiple imputation addressed missing data; Odds Ratio (OR) = 6.71, 95% CI 2-sided [0.86 to 52.14] — The placebo/methotrexate group was the reference category

65. Secondary Outcome: Psoriatic Arthritis Skin Index (PASI) Response at 52 Weeks
Description: as for outcome 62
Time Frame: 52 Weeks
Population: Full Analysis Set (restricted to those with >=3% body surface area affected by psoriasis at baseline)
Measure: Count of Participants; unit: Participants
Arm/Group | Methotrexate | Golimumab & Methotrexate
Number analyzed (Participants) | 8 | 13
Participants | 2 | 6
Statistical Analysis 1: Comparison: Methotrexate vs Golimumab & Methotrexate; Test type: Superiority; p = 0.397, Regression, Logistic; Adjusted for poly/oligoarthritis status (the stratification variable). Multiple imputation addressed missing data; Odds Ratio (OR) = 2.34, 95% CI 2-sided [0.33 to 16.66] — The placebo/methotrexate group was the reference category

66. Secondary Outcome: Ultrasound Imaging Remission at 12 Weeks
Description: Ultrasound Imaging Remission (coded 0=No, 1=Yes) is achieved when all joints and entheses score grey scale<=1 & power Doppler=0.
Time Frame: 12 Weeks
Population: Full Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Methotrexate | Golimumab & Methotrexate
Number analyzed (Participants) | 41 | 43
Participants | 4 | 1
Statistical Analysis 1: Comparison: Methotrexate vs Golimumab & Methotrexate; Test type: Superiority; p = 0.309, Regression, Logistic; Adjusted for poly/oligoarthritis status (the stratification variable). Multiple imputation addressed missing data; Odds Ratio (OR) = 0.33, 95% CI 2-sided [0.04 to 2.83] — The placebo/methotrexate arm was the reference category

67. Secondary Outcome: Ultrasound Imaging Remission at 24 Weeks
Description: as for outcome 66
Time Frame: 24 Weeks
Population: Full Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Methotrexate | Golimumab & Methotrexate
Number analyzed (Participants) | 41 | 43
Participants | 3 | 3
Statistical Analysis 1: Comparison: Methotrexate vs Golimumab & Methotrexate; Test type: Superiority; p = 0.871, Regression, Logistic; Adjusted for poly/oligoarthritis status (the stratification variable). Multiple imputation addressed missing data; Odds Ratio (OR) = 0.87, 95% CI 2-sided [0.17 to 4.60] — The placebo/methotrexate group was the reference category

68. Secondary Outcome: Ultrasound Imaging Remission at 36 Weeks
Description: as for outcome 66
Time Frame: 36 Weeks
Population: Full Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Methotrexate | Golimumab & Methotrexate
Number analyzed (Participants) | 41 | 43
Participants | 2 | 1
Statistical Analysis 1: Comparison: Golimumab & Methotrexate; Test type: Superiority; p = 0.555, Regression, Logistic; Adjusted for poly/oligoarthritis status (the stratification variable). Multiple imputation addressed missing data; Odds Ratio (OR) = 0.48, 95% CI 2-sided [0.04 to 5.52] — The placebo/methotrexate group was the reference category

69. Secondary Outcome: Additional Steroid Received Before 24 Weeks
Description: Participants were eligible for additional steroid at weeks 8 and 12 if they had not achieved a PsARC response; this variable was coded 0=No, 1=Yes.
Time Frame: 12 Weeks
Population: Full Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Methotrexate | Golimumab & Methotrexate
Number analyzed (Participants) | 41 | 43
Participants | 20 | 9
Statistical Analysis 1: Comparison: Methotrexate vs Golimumab & Methotrexate; Test type: Superiority; p = 0.009, Regression, Logistic; Adjusted for poly/oligoarthritis status (the stratification variable). Multiple imputation addressed missing data; Odds Ratio (OR) = 0.28, 95% CI 2-sided [0.11 to 0.72] — The placebo/methotrexate group was the reference category

ADVERSE EVENTS:
Time Frame: 52 Weeks
Description: Determination of AEs was based on the signs or symptoms detected during the physical examination and on clinical evaluation of the participants, and was assessed and recorded at every visit.
  AEs and SAEs were collected from first dose of protocol treatment until week 52. Participants were instructed to report AEs and SAEs during this time period.
Arm/Group | Methotrexate | Golimumab & Methotrexate
All-Cause Mortality (participants affected / at risk) | 0/41 | 0/43
Serious Adverse Events (participants affected / at risk) | 0/41 | 0/43
Other Adverse Events (participants affected / at risk) | 38/41 | 41/43
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Methotrexate (N=41) | Golimumab & Methotrexate (N=43)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Blurred vision (Eye disorders) | 0 (0) | 1 (1)
Cataract (Eye disorders) | 1 (1) | 0 (0)
Dry eye (Eye disorders) | 2 (2) | 3 (3)
Flashing lights (Eye disorders) | 1 (1) | 0 (0)
Glaucoma (Eye disorders) | 0 (0) | 1 (1)
Vitreous hemorrage (Eye disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 2 (3) | 1 (1)
Bloating (Gastrointestinal disorders) | 2 (2) | 0 (0)
Constipation (Gastrointestinal disorders) | 2 (2) | 0 (0)
Dental caries (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 6 (7) | 10 (10)
Dyspepsia (Gastrointestinal disorders) | 2 (2) | 3 (3)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 2 (2) | 0 (0)
Mucositis oral (Gastrointestinal disorders) | 3 (3) | 1 (1)
Nausea (Gastrointestinal disorders) | 11 (14) | 16 (24)
Other: Broken tooth (Gastrointestinal disorders) | 0 (0) | 1 (1)
Other: Fatty infiltration of pancreas (Gastrointestinal disorders) | 1 (1) | 0 (0)
Other: Loose stools (Gastrointestinal disorders) | 1 (1) | 0 (0)
Other: Mouth ulcers (Gastrointestinal disorders) | 2 (2) | 0 (0)
Stomach pain (Gastrointestinal disorders) | 2 (2) | 0 (0)
Vomiting (Gastrointestinal disorders) | 6 (8) | 1 (1)
Fatigue (General disorders) | 3 (3) | 10 (10)
Flu like symptoms (General disorders) | 4 (4) | 2 (2)
Non-cardiac chest pain (General disorders) | 1 (1) | 1 (1)
Other: Fatty liver (Hepatobiliary disorders) | 1 (1) | 0 (0)
Other: Hepatic steatosis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Other: Liver fibrosis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Other: Steatohepatitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Allergic reaction (Immune system disorders) | 1 (1) | 1 (1)
Abdominal Infection (Infections and infestations) | 1 (2) | 0 (0)
Bladder infection (Infections and infestations) | 0 (0) | 1 (1)
Enterocolitis infectious (Infections and infestations) | 0 (0) | 2 (2)
Herpes simplex reactivation (Infections and infestations) | 1 (1) | 0 (0)
Laryngitis (Infections and infestations) | 0 (0) | 1 (1)
Lung infection (Infections and infestations) | 1 (1) | 0 (0)
Mucosal infection (Infections and infestations) | 0 (0) | 3 (4)
Nail infection (Infections and infestations) | 0 (0) | 1 (1)
Other: Genital thrush (Infections and infestations) | 0 (0) | 1 (1)
Otitis externa (Infections and infestations) | 0 (0) | 1 (2)
Papulopustular rash (Infections and infestations) | 1 (1) | 0 (0)
Pharyngitis (Infections and infestations) | 2 (2) | 1 (1)
Shingles (Infections and infestations) | 0 (0) | 1 (1)
Skin infection (Infections and infestations) | 5 (6) | 3 (3)
Soft tissue infection (Infections and infestations) | 2 (2) | 0 (0)
Upper respiratory infection (Infections and infestations) | 12 (13) | 18 (26)
Urinary tract infection (Infections and infestations) | 5 (7) | 0 (0)
Vaginal infection (Infections and infestations) | 0 (0) | 1 (1)
Bruising (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Burn (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Other: Skin injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Other: Spider bite (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Other: Twisted right knee (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Other: Vaccine complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Wrist fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 15 (23) | 21 (35)
Aspartate Aminotransferase increased (Investigations) | 0 (0) | 1 (1)
Blood bilirubin increased (Investigations) | 1 (1) | 1 (2)
Creatinine increased (Investigations) | 1 (1) | 0 (0)
Neutrophil count decreased (Investigations) | 2 (2) | 5 (6)
Other: HBA1C elevated (Investigations) | 1 (1) | 0 (0)
Other: Macrocytosis (Investigations) | 0 (0) | 3 (3)
Other: Vitamin D insufficiency (Investigations) | 7 (8) | 1 (1)
Platelet count decreased (Investigations) | 0 (0) | 3 (3)
Weight gain (Investigations) | 4 (4) | 2 (3)
Weight loss (Investigations) | 0 (0) | 1 (1)
White blood cell decreased (Investigations) | 1 (1) | 3 (3)
Anorexia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Glucose intolerance (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Muscle cramp (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Other: Mass right forearm (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Other: Muscle spasm (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Other: Raynaud's phenomenon (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Other: Trigger finger (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 2 (2) | 3 (3)
Headache (Nervous system disorders) | 3 (3) | 4 (4)
Other: Restless legs syndrome (Nervous system disorders) | 1 (1) | 0 (0)
Paresthesia (Nervous system disorders) | 0 (0) | 1 (1)
Somnolence (Nervous system disorders) | 0 (0) | 2 (2)
Anxiety (Psychiatric disorders) | 0 (0) | 3 (3)
Depression (Psychiatric disorders) | 0 (0) | 3 (3)
Insomnia (Psychiatric disorders) | 0 (0) | 3 (3)
Libido decreased (Psychiatric disorders) | 1 (1) | 0 (0)
Other: Mood swings (Psychiatric disorders) | 1 (1) | 0 (0)
Urinary frequency (Renal and urinary disorders) | 0 (0) | 2 (2)
Dyspareunia (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Erectile Dysfunction (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Irregular menstruation (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Menorrhagia (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Other: Erythematous lesion at the tip of penis, balanitis (dermatologist confirmed) (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Other: High secretion from the breast (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Uterine haemorrhage (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pharyngeal mucositis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (2)
Dyshidrotic eczema (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0)
Other: Contact dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Flushing (Vascular disorders) | 0 (0) | 2 (2)
Hematoma (Vascular disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 3 (4) | 3 (3)
Other: Varicose veins (Vascular disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2022-03-09): https://cdn.clinicaltrials.gov/large-docs/68/NCT04108468/Prot_000.pdf
  • Statistical Analysis Plan (2023-11-17): https://cdn.clinicaltrials.gov/large-docs/68/NCT04108468/SAP_001.pdf